CLINICAL TRIAL: NCT01422941
Title: A PROSPECTIVE, MULTI-CENTER CLINICAL EVALUATION TO ASSESS SAFETY AND PERFORMANCE OF CAVU MEDICAL, INC.'S ATTUNE TUBING WHEN USED WITH NEWLY-IMPLANTED LAPAROSCOPIC ADJUSTABLE GASTRIC BANDS (LAGBs)
Brief Title: Safety and Performance of the CAVU Medical, Inc. Attune Tubing Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cavu Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0271
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2011-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAVU Attune Device (Experimental)
  Interventions: Device: CAVU Attune Device

INTERVENTIONS:
Device: CAVU Attune Device — The CAVU Attune device is used with LAGB.

SUMMARY:
The objectives of this clinical research project are to demonstrate the safety and feasibility of CAVU Medical, Inc.'s Attune Device.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age.
2. The subject has been informed of the nature of the trial and agrees to its provisions.
3. The subject has a pre-implantation BMI within the protocol limits.
4. The subject agrees to the follow-up visit schedule.
5. The subject is a candidate for a LAGB procedure.
6. The subject agrees to comply with specified follow-up evaluations.
7. The subject is willing to fast for 2 hours prior to each adjustment visit.

Exclusion Criteria:

1. The subject is pregnant or is not willing to use an effective method of birth control for the duration of the trial.
2. The subject has a condition that is contraindicated for LAGB procedures.
3. The subject is currently using weight loss medications or supplements.
4. The subject has a concurrent terminal medical condition with a life expectancy of less than 12 months.
5. The subject is currently participating in an investigational drug or another medical device trial.
6. The subject had a previous LAGB procedure.
7. The Investigator believes that the patient has physical or mental conditions that would render trial participation inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The rate of successful placement and filling of the CAVU Medical Attune device without serious device-related adverse events. | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Brancatisano, B Appl Sc, Principal Investigator — Institute of Weight Control
Locations (2):
- Australia (2):
  - Institute of Weight Control, Baulkham Hills, New South Wales
  - St. George Private Hospital, Kogarah, New South Wales